CLINICAL TRIAL: NCT05164718
Title: The Norwegian Exercise in Atrial Fibrillation Trial - An Open-label, Multicenter Randomized Controlled Trial Comparing an eHealth-based Exercise Intervention With Usual Care After 12 Months Follow-up
Brief Title: The Norwegian Exercise in Atrial Fibrillation Trial
Acronym: NEXAF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); UiT The Arctic University of Norway (Other); University Hospital of North Norway (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 213848; 90538300 (Other Grant/Funding Number: Samarbeidsorganet); 315578 (Other Grant/Funding Number: Norwegian Research Council); 22568 (Other Grant/Funding Number: Norwegian Health Association)
Record Dates: First submitted 2021-11-18; First posted 2021-12-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation
Keywords: Exercise therapy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants are not blinded to group allocation. Researchers will be blinded to group allocation when performing statistical analyses. At study completion, a de-identified copy of the data will be extracted for statistical analyses. Information on group allocation will be kept at the Clinical research Unit in Mid-Norway and provided to the research team once a blinded interpretation of the results is finalized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Behavioral: Supervised home-based exercise
- Control group (Other)
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Supervised home-based exercise — 150-300 minutes of moderate intensity activity (55-75% of maximum heart rate in sinus rhythm or RPE 12-13 on the Borg Scale) or 75-150 minutes of vigorous intensity activity (75-90% of maximum heart rate or 14-16 on the Borg Scale) per week, or an equivalent combination of both, according to current general recommendations, including also those with established CVD. To maximize the potential for improvements in cardiorespiratory fitness, we encourage that at least 40-60 minutes per week (i.e. 2 sessions á 20-30 minutes) should be of vigorous intensity.
  Arms: Exercise group
Other: Usual care — Standard management according to usual practice at the respective participating centers, including medical therapy as per guidelines. Prior to randomization all will be provided an ICM (Confirm RX™). The UC group will receive information about general PA recommendations as per guidelines at study enrollment. No further supervision is given.
  Arms: Control group

SUMMARY:
Atrial fibrillation (AF) patients suffer a high symptom burden and reduced quality of life (QoL), high hospitalization rates and few effective treatment options. They have a high burden of cardiovascular risk factors and events. Lifestyle changes and exercise is a cornerstone of management in most chronic cardiac conditions and holds promise in AF, but the evidence is sparse and specific guidelines for exercise do not exist for AF patients. NEXAF is a large-scale multicenter randomized trial to determine the feasibility and effects of exercise on patient-reported and clinical outcomes. All patients will undergo continuous rhythm monitoring, enabling assessment of duration, frequency and total time of AF episodes. The overall aim of the study is to provide documentation for clinical exercise recommendations in AF. The objectives are to examine the effects of a 1-year exercise intervention in AF patients on (i) QoL and symptom burden, (ii) time-in-AF, and peak oxygen uptake, cardiac structure and function, cardiovascular risk factors and use of healthcare resources.

DETAILED DESCRIPTION:
A pre-planned substudy will examine the immediate (24-h to 7 days) effects of vigorous exercise on AF-burden in a subgroup of participants from each arm. Two main outcomes are prespecified: (i) mean time-in-AF measured by an insertable cardiac monitor (ICM) 24 hours after maximal exercise testing at baseline and follow-up compared to mean of the last week before exercise test. (ii) Normal cardiac biomarker response for Troponin and NT-proBNP to acute exercise (0h, 3h, 24h post exercise). Secondary outcomes are mean time-in-AF the consecutive week and post-exercise heart rate variability and number of atrial and ventricular extra systoles at the same time points. Further, changes in post-exercise responses after the intervention (12 months) and the effect on clinical outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosed with paroxysmal or persistent AF in hospital registries
* In sinus rhythm at baseline screening
* Report <75 minutes per week of vigorous and/or <150 minutes of moderate intensity exercise the last three months
* Use a smartphone

Exclusion Criteria:

* Permanent AF or persistent AF with at least one continuous episode lasting ≥3 months the last year
* AF as a complication of acute coronary syndromes, cardiothoracic surgery or infections
* Planned ablation procedure next 12 months or ablated last 6 months without known recurrence
* Unstable coronary heart disease
* De-compensated heart failure
* Left ventricular ejection fraction <40%
* At least moderate to severe mitral or aortic pathology, or aortic aneurysms clinically incompatible with safe exercise
* Moderate to severe chronic obstructive pulmonary disease (GOLD group C+D)
* Ongoing severe cancer or active cancer treatment
* Pacemaker or ICD
* Pregnancy
* Alcohol or drug abuse
* Cognitive or serious psychiatric disease that may impede protocol compliance
* Physical impairments or diseases hindering exercise or making exercise contraindicated
* Resident of nursing home or other institution
* Participation in conflicting research studies (i.e. lifestyle interventions)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life and symptoms | 12 months
  Overall score (0-100) of the 20-item Atrial Fibrillation Effect and Quality of Life (AFEQT) questionnaire. The subscale scores on symptoms, daily activities, and treatment concern, respectively, and the overall score at 6 months, will aid to interpretation as secondary endpoints. Two questions regarding satisfaction with health care providers and treatment are not included in the overall score and will not be collected.
Total time-in-AF(%) | 12 months
  Measured by implantable loop recorder over 12 months

SECONDARY OUTCOMES:
Frequency and duration of AF episodes | 12 months
  Number of recorded AF episodes during follow-up will be calculated from the continuous ILR measurement over the 12 months. We will analyze between group differences (exercise vs. conventional management) in number of continuous AF episodes ≥6min, ≥60min, ≥24h and ≥7 days, respectively, as well as differences in median episode duration.
Frequency and severity of atrial fibrillation symptoms | 6 and 12 months
  Measured by the 16-item AF symptoms and severity checklist. Total score on frequency and severity, respectively, and a subscore of AF-specific symptoms will be analyzed.
Change in peak oxygen uptake (VO2peak) | 12 months
  Measured by ergospirometry pre- and post-intervention
Change in physical and mental dimensions of health | 6 months and 12 months
  The 12 item RAND-12 questionnaire corresponding to eight principal physical and mental health domains. Summarized into two scores; "Physical Health Summary Measure (PCS-physical component score)" and "Mental Health Summary Measure (MCS-mental component score). The EQ-VAS score will ask the patients to simply rate their current health status on a 0-100 scale ranging from "the best health you can imagine" to "the worst health you can imagine".
Change in cardiovascular risk factors | 12 months
  Sum of z-scores of waist, blood pressure, HDL-cholesterol, triglycerides and glucose.
Changes in cardiac volume and dimensions | 12 months
  Echocardiographic indices of left atrial end-systolic volume (crude and indexed to body surface area), left ventricular end-diastolic volume and left atrial end-systolic to left ventricular end-diastolic volume ratio
Incident mortality, cardiovascular events, cardioversions, ablations and total hospitalization | 12 months
  Information about hospitalizations and the discharge diagnoses will be collected by journal review
Safety outcome parameters | 12 months
  Death or unplanned hospitalization summarized per treatment group.
Physical activity level and adherence | 6 and 12 months.
  Self-reported physical activity (PA) will be measured by questionnaire consisting of 3 items (frequency, duration and intensity of regular exercise) in both groups at baseline, 6- and 12 months. Responses of frequency (exercise sessions per week) will be combined with duration of exercise (minutes per session) to estimate weekly minutes of exercise. Minutes of exercise will then be combined with reported intensity (light, moderate, vigorous) to calculate exercise volume and evaluate adherence to the intervention (numbers above and below recommended volume).

OTHER OUTCOMES:
Other changes in cardiac structure and function | 12 months
  Echocardiographic indices of atrial and ventricular structure and function
Change in blood pressure | 12 months
  Change in resting systolic, diastolic and mean arterial blood pressure (diastolic BP + 1/3 x pulse pressure) measured in mmHg at baseline and 12 months.
Change in lipids | 12 months
  Change in HDL-, LDL-, total cholesterol and triglycerides measured in mmol/L at baseline and 12 months.
Change in body weight | 12 months
  Change in body weight measured in kilograms in all participants at baseline and 12 months. Change in fat- and muscle mass in kilograms in a subgroup of participants at baseline and 12 months.
Acute biomarker response to high-intensity exercise | 0, 3 and 24 hours, respectively, after maximal exercise test compared to resting values at baseline and 12 months follow-up
  Level of hs-troponins, NT-proBNP and inflammatory markers pre and post maximal exercise. Biomarker response as predictors of change in AF burden and cardiac remodelling and future events will be evaluated, as well as change in biomarker response post-intervention.
Cognitive function parameters | 12 months
  Measured by a web-based test battery (Memoro)
Usability | 12 months
  Measured by the 10-item system usability scale.
Immediate effects of vigorous exercise on time-in-atrial fibrillation | 0-7 days (daily and cumulative) after maximal test pre- and post-intervention
  Post-exercise time-in-atrial fibrillation (% of day) measured by implantable loop recorder, heart rate and variability and other rhythm parameters (i.e. ventricular and atrial extrasystoles) the following days after a maximal exercise test will be compared to baseline values the preceding days. Echocardiographic predictors of post-exercise AF episodes will be evaluated.
Perceived competence for exercise | 12 months
  Perceived competence will be measured using overall score (4-28, higher score indicates better competence) of the 4-item perceived competence scale (PCS) for regular exercise in both groups at 12 months.
Self-efficacy for exercise | 12 months
  Self-efficacy will be measured using the overall score (9-90, higher score indicates better self-efficacy) of the 9-item Self-Efficacy for Exercise Scale (SEE-EX) in both groups at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Study Director — NTNU, Department of Circulation and Medical Imaging; Rune Wiseth, md phd, Study Director — St Olavs Hospital, Clinic of Cardiology; Bjarne M Ness, phd, Principal Investigator — NTNU, Department of Circulation and Imaging
Locations (3):
- Norway (3):
  - Vestre Viken HF, Drammen
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nes BM, Letnes JM, Johnson KE, Sellevold AB, Byrkjeland R, Brown FP, Follestad T, Dalen H, Wisloff U, Lochen ML, Tveit A, Morseth B, Myrstad M, Loennechen JP; NEXAF consortium; The NEXAF consortium. Effects of 1-year exercise in patients with atrial fibrillation: study protocol for the Norwegian Exercise in Atrial Fibrillation (NEXAF) randomised controlled trial. Open Heart. 2025 Mar 22;12(1):e003077. doi: 10.1136/openhrt-2024-003077. PMID 40122568